CLINICAL TRIAL: NCT05131425
Title: Group Cognitive Behavioral Treatment for Anxiety in Adolescents With ASD and Intellectual Disability: A Randomized Controlled Trial
Brief Title: Facing Your Fears: Adolescents With ASD and Intellectual Disability
Acronym: FYF:ASD/ID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-3142
Record Dates: First submitted 2021-07-08; First posted 2021-11-23 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability; Anxiety; Emotion Regulation
Keywords: autism spectrum disorder; intellectual disability; cognitive behavioral therapy; anxiety; emotion regulation
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Anxiety Disorders; Emotional Regulation | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: The main objective of the current proposal is to conduct an RCT (i.e., treatment group and treatment-as-usual (TAU) control group) to examine the impact of a cognitive behavioral treatment for anxiety in an adolescent sample of Autistic youth with intellectual disability. This clinical trial incorporates random assignment, a control group, and a treatment group. All participants in the TAU control group can crossover and complete the intervention.
Who Masked: Outcomes Assessor
Masking Description: A blinded clinical evaluator will assess outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Intervention (Experimental): The experimental condition is a CBT intervention which focuses on developing 1) emotion regulation skills, 2) somatic management skills individually tailored for sensory and regulatory needs; 3) cognitive strategies such as individualized helpful thoughts and mantras (I can do it); and 4) graded exposure (e.g., facing fears).
  Interventions: Behavioral: Facing Your Fears: ASD/ID
- Treatment as Usual (Other): The TAU condition will serve as the control condition and participants' medication use and outside therapies will be tracked monthly. Following completion of the 16-week wait period, the TAU group will be invited to enroll in FYF:ASD/ID.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Facing Your Fears: ASD/ID — This cognitive behavioral therapy, entitled Facing Your Fears for Adolescents with Autism and Intellectual Disability, is focused on somatic management, helpful cognitive mantras, emotion regulation, and graduated exposure adapted for the cognitive and linguistic needs of an Intellectual Disability population.
  Other Names: Cognitive behavioral therapy
  Arms: Cognitive Behavioral Intervention
Other: Treatment as Usual — The treatment as usual condition is being used in this study as a control condition. The investigators will track what medication and intervention services families are currently receiving.
  Arms: Treatment as Usual

SUMMARY:
Adolescents with ASD and intellectual disability (ID) are a complex and underserved population. Approximately 50% of individuals with ASD/ID experience significant anxiety. Yet, there are very limited mental health care interventions available for this population. Addressing anxiety and building coping skills is particularly important during adolescence as coping skills can support a successful transition to adulthood and family functioning during a difficult developmental period.

The current investigators adapted a cognitive behavioral treatment (CBT) manualized intervention, Facing Your Fears, for adolescents with ASD/ID (FYF:ASD/ID) and completed a pilot study with 23 teens. Preliminary results indicated significant improvements in anxiety and mood symptoms. The proposed study seeks to test whether FYF:ASD/ID is more effective in reducing anxiety than treatment-as-usual (TAU). The investigators propose a Randomized Control Trial (RCT) with 36 adolescents with ASD/ID (12-18 years) randomized to FYF: ASD/ID and 36 adolescents randomized to TAU for 14 weeks. The 36 teens randomized to TAU will then cross-over and complete FYF:ASD/ID. Evaluations will take place at Baseline, Post-Intervention, and 6-month follow-up. Teens in the TAU will have two baseline assessments prior to crossing over to FYF:ASD/ID; both groups will complete a 6-month follow-up assessment after finishing FYF:ASD/ID.

There are three aims for this project: (1) examine the efficacy of FYF: ASD/ID relative to TAU in improving anxiety as measured by parent report and determine if any gains noted in the FYF:ASD/ID are maintained at 6-month follow-up; (2) examine secondary outcomes of anxiety such as how emotion regulation and problem behavior are affected by participation in FYF:ASD/ID; and (3) examine whether adolescents' independent use of CBT skills (as assessed by goal attainment ratings of prompting level required to use strategies) to manage anxiety are increased following participation in FYF:ASD/ID.

DETAILED DESCRIPTION:
Background: Adolescents with ASD and intellectual disability (ID) are a complex and under-served population. Anxiety occurs at higher rates in individuals with ASD/ID (53%) than in ID alone (17%) and may result in physical distress, avoidance of stressful situations, and problem behavior. Further, it frequently contributes to caregivers "taking over" tasks for youth with ID and limiting independence. Parents voice concern about treatment options as the limited available supports often focus on prevention and accommodation of anxiety, rather than on building coping skills. Thus, teens often finish high school with limited coping abilities and consequently experience heightened anxiety in the workplace and poor job retention. Yet, when coping skills are taught early in adolescence, there is an opportunity to practice coping prior to transition, leading to better employment rates, decreased clinical service use, and increased long-term wages. Addressing anxiety and building coping skills for teens with ASD/ID is of critical importance as these are per-requisite skills for successful transition to adulthood.

Intervention: A significant treatment barrier for teens with ASD/ID is the lack of evidence based, manualized interventions for this population. This is due, in part, because youth with ASD/ID have typically been excluded from intervention research trials examining the effectiveness of best practice treatments such as cognitive behavioral therapy (CBT). Recent research adapting CBT to meet the cognitive, social, and behavioral needs of this population have yielded promising results and challenge the paradigm that individuals with ID are not able to access cognitive and emotion regulation strategies. The research team for the present study adapted a CBT manualized intervention, Facing Your Fears, for adolescents with ASD/ID (FYF:ASD/ID) and completed a pilot study with 23 teens. Preliminary outcome measures indicated significant improvements in anxiety and mood symptoms.

Objective: The current study seeks to test whether FYF:ASD/ID, an adapted CBT intervention for teens with ASD/ID, is more effective in reducing anxiety than treatment-as-usual (TAU).

Study Design: The investigators will use a Randomized Control Trial (RCT) with 36 adolescents with ASD/ID (12-18 years) randomized to FYF: ASD/ID and 36 adolescents randomized to TAU for 14 weeks. The 36 teens randomized to TAU will then cross-over and complete FYF:ASD/ID. Evaluations will take place at Baseline, Post-Intervention, and 6-month follow-up. Teens in the TAU will have two baseline assessments prior to crossing over to FYF:ASD/ID; both groups will complete a 6-month follow-up assessment after finishing FYF:ASD/ID.

Specific Aims: Three aims are proposed: (1) examine the efficacy of FYF: ASD/ID relative to TAU in improving anxiety as measured by parent report and determine if gains are maintained at 6-month follow-up; (2) examine secondary outcomes of anxiety such as how emotion regulation and problem behavior are affected by participation in FYF:ASD/ID; and (3) examine whether adolescents' independent use of CBT skills (as assessed by goal attainment ratings of prompting level required to use strategies) to manage anxiety are increased following participation in FYF:ASD/ID.

Impact: The present study would represent the first RCT of a CBT intervention for adolescents with ASD/ID, a critical step toward establishing an evidence base for anxiety treatment for this underserved and vulnerable population.

Translatability: It is necessary to close the gap in the availability of anxiety interventions and ensure effective mental health care for all individuals on the spectrum. Completing a well-designed RCT that incorporates random assignment, a control group, and careful measurement of anxiety is a critical next step in evaluating the effectiveness of this CBT treatment and supporting the study of interventions that can contribute to positive coping skills that allow teens to access time limited transition services and optimize outcome.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age between 12-18 years
* A confirmed diagnosis of ASD, as based on a score above ASD cutoff on the Autism Diagnostic Observation Schedule-Second Edition and DSM-5 clinical evaluation
* Cognitive and adaptive behavior abilities in the ID range as determined by a Brief IQ standard score between 40 - 70 on the Stanford Binet-Fifth Edition (SB-5) and a Total Adaptive Composite below 70 on the Adaptive Behavior Assessment System, 3rd Edition (ABAS-3)
* Clinically significant symptoms of anxiety, defined by clinically significant anxiety elevations on the ADAMS and meeting diagnostic criteria for at least one anxiety diagnosis on the Anxiety Disorders Interview Schedule: Autism Addendum (ADIS:ASA)

Exclusion Criteria:

* A primary mental health diagnosis of a non-anxiety psychiatric condition such as a thought disorder, as determined following administration of the ADIS:ASA, thus suggesting that a different treatment approach is merited
* A raw score above 18 on the Irritability sub-scale of the Aberrant Behavior Checklist-Community (ABC-C), indicating problem behavior is 1.5-2 SD above the mean for youth with ID within this age range, thus suggesting a group treatment may not be appropriate
* Inability of families to attend at least 11 of 14 sessions

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in number of anxiety diagnoses as measured by the Anxiety Disorders Interview Schedule: Autism Addendum (ADIS:ASA) | Baseline (i.e., within 6 weeks' start of the treatment or TAU condition), Post treatment (i.e., within 6 weeks of the completion of the14-week treatment or TAU condition), and follow-up (six months following the completion of the treatment condition)
  The ADIS:ASA is a semi-structured clinical interview completed with a parent that assesses anxiety diagnoses in children and adolescents with ASD. This measure provides a total number of anxiety diagnoses for a child. The interview will be administered and anxiety diagnoses recorded at the following time points: Baseline (i.e., within 6 weeks' start of the treatment or TA condition), Post treatment (i.e., within 6 weeks of the completion of the14-week treatment or TAU condition), and follow-up (six months following the completion of the treatment condition). Change in the total number of anxiety diagnoses that a child meets diagnostic criteria for on the ADIS:ASA will be calculated across the aforementioned time points.
Change in the Clinical Global Improvement-Severity score as derived by the Anxiety Disorders Interview Schedule: Autism Addendum (ADIS:ASA) | Baseline (i.e., within 6 weeks' start of the treatment or TAU condition), Post treatment (i.e., within 6 weeks of the completion of the14-week treatment or TAU condition), and follow-up (six months following the completion of the treatment condition)
  Clinical Global Improvement-severity (CGI-S) scores are derived from the ADIS:ASA. The CGI-S is a summary rating (i.e., likert scale of 1 to 7 with 7 indicating very severe) indicating the extent to which the teen's anxiety symptoms assessed via the ADIS:ASA impact daily functioning. To calculate change in anxiety severity, the CGI-S ratings are calculated at baseline (i.e., 6 weeks prior to the start of the 14-week TAU condition of intervention condition), post-treatment (i.e., within 6 weeks of the end of the completion of the 14-week TAU condition and intervention group conditions) and at follow-up (i.e., 6 months following the completion of the 14-week TAU intervention group). Change in CGI-S ratings across these time points are calculated.

SECONDARY OUTCOMES:
Change in the Reactivity subscale as assessed by the Emotion Dysregulation Inventory (EDI) | Baseline (i.e., within 6 weeks' start of the treatment or TAU condition), Post treatment (i.e., within 6 weeks of the completion of the14-week treatment or TAU condition), and follow-up (six months following the completion of the treatment condition)
  The EDI is a parent report measure of emotion dysregulation in youth with ASD. Items are rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very severe). The Reactivity sub-scale contains 7-items. Possible scores on the Reactivity sub-scale could range from 7 to 35, with higher scores indicating a worse outcome. To calculate change in Reactivity the total score on the sub-scale is calculated at baseline (i.e., 6 weeks prior to the start of the 14-week TAU condition of intervention condition), post-treatment (i.e., within 6 weeks of the end of the completion of the 14-week TAU condition and intervention group conditions) and at follow-up (i.e., 6 months following the completion of the 14-week TAU intervention group).
Change in the Dysphoria subscale as assessed by the Emotion Dysregulation Inventory (EDI) | Baseline (i.e., within 6 weeks' start of the treatment or TAU condition), Post treatment (i.e., within 6 weeks of the completion of the14-week treatment or TAU condition), and follow-up (six months following the completion of the treatment condition)
  The EDI is a parent report measure of emotion dysregulation in youth with ASD. Items are rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very severe). The Dysphoria subscale contains 6-items. Possible scores on the Reactivity subscale could range from 6 to 30, with higher scores indicating a worse outcome. To assess change in Dysphoria, the total score on the Dysphoria subscale is calculated at baseline (i.e., 6 weeks prior to the start of the 14-week TAU condition of intervention condition), post-treatment (i.e., within 6 weeks of the end of the completion of the 14-week TAU condition and intervention group conditions) and at follow-up (i.e., 6 months following the completion of the 14-week TAU intervention group). Change is assessed across these time points.
Change in problem behavior as assessed by the The Aberrant Behavior Checklist-Community (ABC-C) | Baseline (i.e., within 6 weeks' start of the treatment or TAU condition), Post treatment (i.e., within 6 weeks of the completion of the14-week treatment or TAU condition), and follow-up (six months following the completion of the treatment condition)
  The ABC-C is a 58-item parent report questionnaire that evaluates the presence and severity of problem behavior across five sub-scales: Irritability, Lethargy/Social Withdrawal, Stereotypic Behavior, Hyperactivity/Noncompliance sub-scales, and Inappropriate Speech. Each item is rated on a scale of 0-3 with 0 being "not at all a problem" and 3 being "the problem is severe in degree." Total problem behavior raw scores across the five sub-scales range from 0-174.To assess change in problem behavior, the total raw score is calculated at baseline (i.e., 6 weeks prior to the start of the 14-week TAU condition of intervention condition), post-treatment (i.e., within 6 weeks of the end of the completion of the 14-week TAU condition and intervention group conditions) and at follow-up (i.e., 6 months following the completion of the 14-week TAU intervention group). Change is assessed across these time points.

OTHER OUTCOMES:
Exploratory Aim: Exploratory analyses will be conducted to evaluate the effect of treatment participation on teens' independent use of somatic management, emotion regulation, and cognitive strategies using goal attainment scaling (e.g., GAS) | Baseline (i.e., within 6 weeks' start of the treatment or TAU condition), Post treatment (i.e., within 6 weeks of the completion of the14-week treatment or TAU condition), and follow-up (six months following the completion of the treatment condition)
  Teens use of somatic management, emotion regulation and cognitive strategies is assessed by a clinician via the CBT goal attainment scale interview. Scores from 0-4 are established for each participant based on outlined criteria for strategy use (0 indicates extremely limit skills and high dependence on others to use skills, 4 indicates independent use of skills, low dependence on others to use skills). Ratings are calculated at baseline (i.e., 6 weeks prior to the start of the 14-week TAU condition of intervention condition), post-treatment (i.e., within 6 weeks of the end of the completion of the 14-week TAU condition and intervention group conditions) and at follow-up (i.e., 6 months following the completion of the 14-week TAU intervention group). Change is assessed across these time points. Within-subject changes from baseline to post-treatment and follow-up on GAS will be evaluated using mixed model analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey D Blakeley-Smith, Ph.d., Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blakeley-Smith A, Meyer AT, Boles RE, Reaven J. Group Cognitive Behavioural Treatment for Anxiety in Autistic Adolescents with Intellectual Disability: A Pilot and Feasibility Study. J Appl Res Intellect Disabil. 2021 May;34(3):777-788. doi: 10.1111/jar.12854. Epub 2021 Jan 6. PMID 33410240
- [Background] Bakken TL, Helverschou SB, Eilertsen DE, Heggelund T, Myrbakk E, Martinsen H. Psychiatric disorders in adolescents and adults with autism and intellectual disability: a representative study in one county in Norway. Res Dev Disabil. 2010 Nov-Dec;31(6):1669-77. doi: 10.1016/j.ridd.2010.04.009. Epub 2010 May 20. PMID 20493660
- [Background] Moskowitz LJ, Mulder E, Walsh CE, McLaughlin DM, Zarcone JR, Proudfit GH, Carr EG. A multimethod assessment of anxiety and problem behavior in children with autism spectrum disorders and intellectual disability. Am J Intellect Dev Disabil. 2013 Nov;118(6):419-34. doi: 10.1352/1944.7558.118.6.419. PMID 24432856
- [Background] Sandjojo J, Gebhardt WA, Zedlitz AMEE, Hoekman J, Dusseldorp E, den Haan JA, Evers AWM. Development of the Leiden Independence Questionnaire for Support Staff: a measure of staff behaviour regarding promoting independence of people with intellectual disabilities. J Intellect Disabil Res. 2019 Apr;63(4):286-297. doi: 10.1111/jir.12574. Epub 2018 Dec 5. PMID 30515912
- [Background] O'Nions E, Happe F, Evers K, Boonen H, Noens I. How do Parents Manage Irritability, Challenging Behaviour, Non-Compliance and Anxiety in Children with Autism Spectrum Disorders? A Meta-Synthesis. J Autism Dev Disord. 2018 Apr;48(4):1272-1286. doi: 10.1007/s10803-017-3361-4. PMID 29222612
- [Background] Reaven J, Blakeley-Smith A, Nichols S, & Hepburn, S. (2011). Facing Your Fears: Group Therapy for Managing Anxiety in Children with High-Functioning Autism Spectrum Disorders. Baltimore, MD: Paul Brookes Publishing
- [Background] Hurlbutt K, Chalmers L. Employment and Adults With Asperger Syndrome. Focus on Autism and Other Developmental Disabilities. 2004;19(4):215-222. doi:10.1177/10883576040190040301
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985 Mar;89(5):485-91. PMID 3993694
- [Background] Esbensen AJ, Rojahn J, Aman MG, Ruedrich S. Reliability and validity of an assessment instrument for anxiety, depression, and mood among individuals with mental retardation. J Autism Dev Disord. 2003 Dec;33(6):617-29. doi: 10.1023/b:jadd.0000005999.27178.55. PMID 14714931
- [Background] Vereenooghe L, Flynn S, Hastings RP, Adams D, Chauhan U, Cooper SA, Gore N, Hatton C, Hood K, Jahoda A, Langdon PE, McNamara R, Oliver C, Roy A, Totsika V, Waite J. Interventions for mental health problems in children and adults with severe intellectual disabilities: a systematic review. BMJ Open. 2018 Jun 19;8(6):e021911. doi: 10.1136/bmjopen-2018-021911. PMID 29921688

DOCUMENTS (1):
  • Informed Consent Form (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT05131425/ICF_000.pdf